CLINICAL TRIAL: NCT04895072
Title: Effect of Injection Rate on the Block Sensory Level in the Erector Spine Plane Block
Brief Title: Injection Rate and Erector Spinae Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4/5
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Breast Surgery
Keywords: Erector spinae plane (ESP) block; Postoperative Pain; Breast Surgery
MeSH Terms: conditions — Pain, Postoperative; Bites and Stings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (Active Comparator): standard injection rate will be applied
  Interventions: Procedure: Standard group
- Long group (Active Comparator): long injection rate will be applied
  Interventions: Procedure: Long group

INTERVENTIONS:
Procedure: Standard group — Ultrasound-guided ESP block with 20 mL %0.375 bupivacaine will be administered at a standard injection rate.
  Arms: Standard group
Procedure: Long group — Ultrasound-guided ESP block with 20 mL %0.375 bupivacaine will be administered at a long injection rate.
  Arms: Long group

SUMMARY:
To evaluate the effect of injection rate on the block sensory level in the ESP block.

DETAILED DESCRIPTION:
Many women experience severe acute postoperative pain after breast cancer surgery. Regional techniques are frequently used as a part of multimodal analgesia in breast surgery. Ultrasound-guided erector spinae plane (ESP) block is a preferred method to reduce the postoperative opioid requirement for postoperative pain management. In this study, we aimed to evaluate the effect of injection rate on the block sensory level in the ESP block.

ELIGIBILITY:
Inclusion Criteria:

* aged between eighteen and sixty-five
* ASA I-III
* undergo elective breast cancer surgery

Exclusion Criteria:

* under 18 years of age or over 65 years of age
* ASA IV and above
* declined to give written informed consent
* contraindications of peripheral blocks or local anesthetic infiltration
* history of allergy against local anesthetics
* chronic pain history
* history of hepatic, neuromuscular, cardiac and/or renal failure
* infection at the injection site

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Block sensory level | 12 hours
  Number (average) of dermatomes with sensory block with pinprick and cold methods after the ESP block

SECONDARY OUTCOMES:
Postoperative tramadol consumption | 24 hours
  Postoperative tramadol consumption will be recorded at 24 hours
Assesment of postoperative analgesia | 24 hours
  Post operative pain scores will be assessed using a numerical rating scala (NRS) (from 0=no pain, to10= worst pain imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Arzu Karaveli, Principal Investigator — Antalya TRH
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barrios A, Camelo J, Gomez J, Forero M, Peng PWH, Visbal K, Cadavid A. Evaluation of Sensory Mapping of Erector Spinae Plane Block. Pain Physician. 2020 Jun;23(3):E289-E296. PMID 32517405